CLINICAL TRIAL: NCT06698263
Title: 13-cis Retinoic Acid (Isotretinoin) and Sperm Production
Acronym: ARESPERM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7345; 2024-519644-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Men with Infertility
MeSH Terms: interventions — Isotretinoin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isotretinoin (Experimental): Isotretinoin (40 mg) orally, once per week for 20 weeks
  Interventions: Drug: Isotretinoin
- control group (Placebo Comparator): Placebo identical in appearance and administration schedule.
  Interventions: Drug: Control group (placebo)

INTERVENTIONS:
Drug: Isotretinoin — ARESPERM is a multicenter, randomized, double-blind, placebo-controlled study that assesses whether a weekly dose of isotretinoin can stimulate spermatogenesis in men with oligozoospermia. The study hypothesizes that isotretinoin can trigger the differentiation of spermatogonial cells, leading to improved sperm production.
  Arms: Isotretinoin
Drug: Control group (placebo) — placebo administration
  Arms: control group

SUMMARY:
This study aims to evaluate the effectiveness of weekly administration of isotretinoin (40 mg) in increasing sperm production in men with oligozoospermia, a condition characterized by a low sperm count. Participants will be randomized into two groups: one receiving isotretinoin and the other a placebo. The primary outcome will be the change in sperm production over 20 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be infertile men (no pregnancy with partner with normal cycles and normal hysterosalpingogram despite >1 year of unprotected intercourse).
* Abnormal sperm analyses with a total, motile sperm count of less than 10 million sperm as assessed by semen analysis on two occasions separated by one week.
* Male patients aged 21-55 years
* Affiliation with a social security system
* Ability to provide informed consent

Exclusion Criteria:

* -Men participating in another clinical trial
* Clinically significant abnormal findings at screening
* Known genetic infertility (e.g. Klinefelter syndrome or Y-chromosome microdeletions),
* Hypogonadotropic hypogonadism (that might respond to gonadotropin injections),
* Severe mental health problems requiring medications
* Current therapy with retinoic acid (e.g. Accutane) or vitamin A.
* History of psychiatric disorders (e.g., depression, suicidal tendencies).
* Abnormal serum chemistry values according to local laboratory normal values which indicate liver or kidney dysfunction.
* Men currently receiving tetracycline containing medications
* Men who have used isotretinoin within eight weeks of the start of dosing
* Men with elevated serum triglycerides

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — just man
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Millions of Sperm Per Ejaculate | Day 0
  Concentration calculation of Millions of sperm per ejaculate in men treated with 13-cis retinoic acid
Millions of Sperm Per Ejaculate | Months 2
  Concentration calculation of Millions of sperm per ejaculate in men treated with 13-cis retinoic acid
Millions of Sperm Per Ejaculate | Months 5
  Concentration calculation of Millions of sperm per ejaculate in men treated with 13-cis retinoic acid
Millions of Sperm Per Ejaculate | Months 12
  Concentration calculation of Millions of sperm per ejaculate in men treated with 13-cis retinoic acid
Millions of Sperm Per Ejaculate | Months 24
  Concentration calculation of Millions of sperm per ejaculate in men treated with 13-cis retinoic acid

CONTACTS AND LOCATIONS:
Locations (1):
- CECOS Alsace Strasbourg, Schiltigheim, France

IPD SHARING:
Plan to Share IPD: No